CLINICAL TRIAL: NCT05179772
Title: Olanzapine Augmentation of Buprenorphine-naloxone Treatment in OUD Patients With Comorbid Symptoms of Serious Mental Illness (SMI): A Prospective Open-label Single-arm 9-week Study
Brief Title: Olanzapine in OUD Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: NIDA has advised us to terminate this protocol due to the difficulties in finding appropriate subjects.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 850369
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olanzapine (Experimental): Everyone in the study is being given Olanzapine (open label)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine (2.5 mg to 20 mg)

SUMMARY:
This study is designed to examine whether olanzapine (2.5 to 20mg/day) impacts opioid use in patients with opioid use disorder and comorbid SMI symptoms who are taking buprenorphine-naloxone. The specified outcomes (e.g., illicit opioid use, other drug use, sleep, MAT adherence, withdrawal and craving, thought and mood disorder symptoms) on olanzapine will be examined within-subjects for change (improvement) across the trial.

Approximately 48 subjects will be enrolled. After enrollment, subjects will complete safety and baseline assessments and will be assigned open-label to 9-weeks olanzapine. Olanzapine will then be tapered over a 1-week period (or maintained if clinically indicated). Urines will be collected 2x/week throughout.

The study has 4 distinct phases: 1) Screening (approx. 1-2 wks); 2) Baseline and Medication Initiation Visit (1 visit; includes safety, baseline and phenotyping measures, study medication dispensed) 3) Outpatient treatment (9 wks; 2 visits/wk, includes daily olanzapine and daily buprenorphine-naloxone (through the participants usual community treatment site and on-medication phenotyping measures); 4) Follow-up visit (1 wk after last dose of study medication).

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for opioid use disorder
* have symptoms of SMI
* on stable dose of buprenorphine-naloxone
* females must either be of non-child bearing potential or on highly-effective contraception

Exclusion Criteria:

* abnormal ECG
* cocaine, alcohol, psychoactive use disorders
* metabolic syndrome or diabetes 1 and 2
* history of seizures
* stable regimen of an antipsychotic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in illicit opioid use | weeks 3-8
  To examine whether adjunctive olanzapine (on top of buprenorphine-naloxone) changes illicit opioid use, indexed by Urine Drug Screens (UDS), in participants with OUD and symptoms of SMI.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kampman, MD, Principal Investigator — University of Pennsylvania; Anna Rose Childress, PhD, Principal Investigator — University of Pennsylvania; Gerard Moeller, MD, Principal Investigator — Virgina Commonwealth University; Albert Arias, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia